CLINICAL TRIAL: NCT04589533
Title: MANAGEMENT OF PATIENTS WITH TYPE 2 DIABETES MELLITUS HOSPITALIZED IN INTERNAL MEDICINE UNITS: A Multicenter Study Before & After Educational Program, With Cluster Randomization (MINDER Study)
Brief Title: MANAGEMENT OF PATIENTS WITH TYPE 2 DIABETES MELLITUS HOSPITALIZED IN INTERNAL MEDICINE UNITS (MINDER Study)
Acronym: MINDER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: FADOI.01.2020
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EDUCATIONAL PROGRAM GROUP: This group will receive an educational program based . This group, as the other group, during phase 1 and phase 3, will review the medical records of the last 40 patients (for each phase) with known T2DM and hospitalized for any cause.
  Interventions: Other: educational program
- CONTROL GROUP: Control group will not receive educational program. This group, as the other group, during phase 1 and phase 3, will review the medical records of the last 40 patients (for each phase) with known T2DM and hospitalized for any cause.

INTERVENTIONS:
Other: educational program — The educational program will be based on: a outreach visit (a 3-h face-to-face meeting between a trained diabetes specialist from outside the Center and the staff of the Center itself) and a distance learning (FAD).The educational programme will be focused on current Diabetes Guidelines recommendations and based on possible deviations from the best clinical practice observed during phase1
  Groups: EDUCATIONAL PROGRAM GROUP

SUMMARY:
This is a national multicenter study that involves 54 Internal Medicine Units throughout Italy. It is designed as a replicate of two cross-sectional surveys interspersed with an educational program. The study is composed by three steps. Phase 1 concerns a retrospective data collection pertaining to patients with known diagnosis of T2DM. In phase 2 an educational training (focused on current Diabetes Guidelines recommendations and based on possible deviations from the best clinical practice observed during phase1) will be conducted in 36 randomized centres out of the 54 ones enrolled (cluster randomization). The ratio 2:1 has been selected in order to offer to the majority of Centres the opportunity to undergo a program of training and maximize the potential positive effect of the educational program on patient management. Randomization will be performed at the beginning of the study. Centres will be selected according to their ability to prescribe all classes of antidiabetic drugs. Phase 3 will occur around 6 months after the training and concerns a new data collection mirroring the previous one. In the phase 1, as well as in the phase 3, the data collection will be based on the review of the medical records of the last 40 consecutive patients with T2DM hospitalized in each Centre of Internal Medicine (in total, 80 patients for each Centre). After a period of 6 months from the hospitalization, a phone call follow up will be performed to know the clinical status of the patient enrolled, if he/she has been re-hospitalized after the index admission and current diabetes treatment.

DETAILED DESCRIPTION:
During phase 1 and phase 3, each Center will review the medical records of the last 40 patients (for each phase) with known T2DM and hospitalized for any cause. Therefore, being the data collection retrospective, patients will be managed according to routine clinical practice. During phase 2, 36 randomized centers, out of the 54 ones enrolled, will receive an educational intervention based on outreach visit (EOV), a 3-h face-to-face meeting between a trained diabetes specialist from outside the Center and the staff of the Center itself. This method was selected being considered as one of the most effective to modify professional practice and improve health care outcomes. In addition, at least 50% of the physicians who are part of the staff of the Center will receive distance learning (FAD). The contents of the educational program will be defined by the study Steering Committee, on the basis of guidelines, and possible deviations from the best medical practice detected during phase 1. In order to minimize the "awareness bias" (i.e. the possibility that participation to the project significantly influence clinical attitudes in phase 3), only one physician of the Centers of the "Control" group (not receiving EOV) will be made aware of the study design and procedures, and he/she will be eventually supported in the study data collection by nurses, or physicians who do not have the possibility of prescribing, in particular regarding the new categories of antidiabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Known diagnosis of type-2 diabetes
3. Informed Consent

Exclusion Criteria:

1. Current treatment with insulin
2. Patients treated with rapid acting insulin during the hospitalization
3. Patients hospitalized for less than 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Internal Medicine and with known diagnosis of diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 4320 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Variation in fasting glycemia between the two groups of Centres during phase 3 of the study | 18 months
  The primary measure will be the variation in fasting glycemia (i.e. calculated by the difference between the fasting glicemia measured ad the admission and the fasting glicemia measured at the hospital discharge) during hospitalization between the two groups of Centres (those receiving and not receiving the educational program) during phase 3 of the study

SECONDARY OUTCOMES:
Variation in fasting glycemia during hospitalization between the phase 1 and phase 3 | 18 months
  To evaluate the variation in fasting glycemia (i.e. calculated by the difference between the fasting glicemia measured ad the admission and the fasting glicemia measured at the hospital discharge) during hospitalization between the phase 1 and phase 3 in the two groups of Centres (those receiving and not receiving the educational program)
Description of characteristics of patients with T2DM hospitalized in Internal Medicine | 18 months
  To describe the characteristics of patients with T2DM hospitalized in Internal Medicine and their treatment

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA FONTANELLA, Study Director — FADOI FOUNDATION
Locations (6):
- Italy (6):
  - Azienda Toscana Nord Ovest, Cecina, Cecina
  - Po Nord "S. Maria Goretti", Latina
  - ASST Sette Laghi, Ospedale Confalonieri di Luino, Luino
  - Ospedale Fatebenefratelli, Napoli
  - Usl Toscana Sud Est, Petruccioli, Pitigliano
  - Presidio di Passirana ASST RHODENSE, Rho

IPD SHARING:
Plan to Share IPD: No